CLINICAL TRIAL: NCT00176969
Title: Perifollicular Nerves in Alopecia Areata: Response to Topical Capsaicin
Brief Title: Response of Topical Capsaicin in Alopecia Areata
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9707M00122
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capsaicin

SUMMARY:
It has been postulated that Alopecia Areata (AA) is, at least in part, a neurologically mediated disease. Research supporting this theory includes the finding that nerves surrounding the hair follicles are collapsed. We want to take this research a step further and show that not only are these perifollicular nerves collapsed, but that their function is also impaired.

DETAILED DESCRIPTION:
To assess the function of perifollicular scalp nerves in AA we will look at the response of these nerves to the topical medication capsaicin. Under normal circumstances topical capsaicin is known to target nerves in the peripheral nervous system causing short-term release of the neuropeptide Substance P (SP) as well as long-term transient depletion of SP. We expect the AA patients will respond abnormally to topical capsaicin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have alopecia totalis or universalis.
* Be in good health.
* Not be taking any medications including topical medications
* Be 18 years or older.
* Be willing to apply study medication or vehicle as directed, comply with instructions and commit to follow-up visits.
* Not have had hair chemically treated (including colored hair, permed hair, etc) within the month prior to the study.

Exclusion Criteria:

* Absence of extensive alopecia areata.
* People not in good health.
* People taking medications.
* Allergies to capsaicin.
* Presence of irritated or visibly inflamed scalp.
* Having had hair chemically treated (including colored hair, permed hair, etc.) within the month prior to study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1997-08; Study Completion 2000-06

PRIMARY OUTCOMES:
Topical capsaicin will quantitatively decrease the amount of Substance P in the scalp of AA patients.

SECONDARY OUTCOMES:
The scalps of AA patients may be less sensitive to stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Marna Ericson, Ph D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States